CLINICAL TRIAL: NCT05348863
Title: SPARK: Smart Phone App for Gestational Diabetes Patients Supporting Key Lifestyle Behaviors and Glucose Control
Brief Title: SPARK- a Digital Platform to Improve Self-management of Gestational Diabetes
Acronym: SPARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Östergötland (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Marie Löf, docent, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-03093
Record Dates: First submitted 2022-04-13; First posted 2022-04-27 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPARK app (Experimental): Access to the SPARK app which will provide support for a healthier diet and increased physical activity as well as daily monitoring of blood glucose levels.
  Interventions: Behavioral: SPARK
- Control arm (No Intervention): Standard care i.e., the routine treatment program for GDM delivered by the care provider.

INTERVENTIONS:
Behavioral: SPARK — The SPARK digital platform provides support to the patient (shown as an app) as well as provides the possibility for the health care provider to review and give feedback on blood glucose levels through the care giver interface of the platform.
  Arms: SPARK app

SUMMARY:
Gestational diabetes mellitus (GDM) is an increasing public health challenge. Innovative, effective and scalable lifestyle interventions to support women with GDM to manage their disease and to prevent adverse obstetric and neonatal outcomes as well as later morbidity are requested.The aim of this project is to evaluate whether a novel, mobile health (mHealth) platform (SPARK) can improve self-management of GDM and prevent adverse maternal and offspring outcomes. SPARK is a multi-centre randomised controlled trial recruiting women diagnosed with GDM in South Eastern Sweden. Women will be randomised to the control or intervention group. All women will receive standard care. The intervention group will also receive support through the SPARK platform for healthy eating, physical activity and glycaemic control. Pregnancy outcomes are glycaemic control (primary), diet, physical activity, metabolic and inflammatory biomarkers in gestational week 36-37 as well as adverse obstetric and neonatal outcomes. Secondary outcomes also include cardiometabolic risk, physical activity and healthy eating behaviours one-year postpartum.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of GDM detected by oral glucose tolerance test in accordance with the World Health Organization guidelines

Exclusion Criteria:

* known pre-pregnancy diabetes
* twin pregnancy
* <18 years of age
* severe co-morbidities that would limit participation or a previously diagnosed severe psychiatric illness.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Glucose control | At the end of the intervention in gestational weeks 36-37
  Time in Range percent of time for glucose levels within clinical target levels using continous glucose monitoring
HbA1c | At the end of the intervention in gestational weeks 36-37
  Glycosylated hemoglobulin

SECONDARY OUTCOMES:
Diet intake quality using three dietary recalls by means of the Riksmaten Flex method | At the end of the intervention in gestational weeks 36-37
  Diet intake quality will be assessed using three 24 hour dietary recalls by means of the Riksmaten Flex web-based dietary recall method.
Physical activity using accelerometry | At the end of the intervention in gestational weeks 36-37
  Time spent on physical activity at different levels (sedentary, light, moderate, vigorous) in minutes per day will be assessed using accelerometry collected during 7 days
Incidence of pre-eclampsia | Up to delivery
  Diagnosis of pre-eclampsia
Incidence of Caesarean sections | Up to delivery
  Delivery by caesarean sections
Incidence of pregnancy induced hypertension | Up to delivery
  Diagnosis of pregnancy induced hypertension
Metformin/insulin treatment | Up to delivery
  Introduction of metformin/insulin treatment
Preterm birth | Up to delivery
  Delivery before 37 completed weeks
Gestational weight gain | From pre-prepregnancy up to 40 weeks of gestation
  Increase in body weight during pregnancy
Infant birth weight | At birth
  Infant birth weight in grams
Infant birth length | At birth
  Infant birth length in centimetres
Infant Apgar score | At birth
  Infant Apgar score at 1, 5 and 10 min
Incidence of large-for gestational-age infant | At birth
  Birth weight >90th percentile for gestational age and gender
Infant shoulder dystocia | At birth
  Incidence of infant shoulder dystocia
Infant hypoglycaemia | At birth
  Incidence of infant hypoglycaemia
Glucose control | From inclusion (baseline) to end of intervention in gestational week 36-37
  Adherence to protocol for daily glucose monitoring (four times per day)
Glycaemic variability I | At the end of the intervention in gestational week 36-37
  Coefficient of variation for glucose excursion over 24 hrs using continous glucose monitoring
Glycaemic variability II | At the end of the intervention in gestational week 36-37
  Mean for glucose excursion over 24 hrs using continous glucose monitoring
Delivery complications | At delivery
  Induction of delivery (yes or no), vacuum extraction (yes or no, epidural anesthesia (yes or no)
Hospital stay | The first week post partum
  Hospital stay (duration from admission of delivery to discharge) including neonatal care
Glucose- insulin treatment during delivery | During delivery
  Incidence of glucose- insulin treatment during delivery
Metabolic and inflammatory biomarkers I | At gestational weeks 36-37
  Maternal levels of Insulin-like Growth Factor I in serum
Metabolic and inflammatory biomarkers II | At gestational weeks 36-37
  Maternal levels of Insulin-like Growth Factor I binding proteins in serum
Metabolic and inflammatory biomarkers III | At gestational week 36-37
  Maternal levels of copeptin in serum
Metabolic and inflammatory biomarkers IV | At gestational week 36-37
  Maternal levels of leptin in serum
Metabolic and inflammatory biomarkers V | At gestational week 36-37
  Maternal levels of midregion pro-adrenomedullin (MR-proANP) in serum
Maternal cardiometabolic risk profile | One year post partum
  A maternal cardiometabolic risk profile score one year post partum will be calculated using information on triglycerides and high-density cholesterol in serum, waist circumference, blood glucose as well as the systolic and diastolic blood pressure.
Diet intake quality using three dietary recalls by means of the Riksmaten Flex method | One year post partum
  Diet intake quality will be assessed using three 24 hour dietary recalls by means of the Riksmaten Flex web-based dietary recall method.
Physical activity using accelerometry | One year post partum
  Time spent on physical activity at different levels (sedentary, light, moderate, vigorous)
Metabolic and inflammatory biomarkers VI | At gestational week 36-37
  Maternal levels of midregion pro-atrial natriuretic peptide (MR-proADM) in serum
Glycaemic variability III | Full intervention period (up to 3 months)
  Glucose levels using glucose meter (capillary sampling)
Microvascular function I | One year post partum
  Oxygen saturation using PeriFlux6000 Enhanced Perfusion and Oxygen Saturation
Microvascular function II | One year post partum
  Total speed perfusion using PeriFlux6000 Enhanced Perfusion and Oxygen Saturation

CONTACTS AND LOCATIONS:
Overall Officials: Marie Löf, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Maternity health care, Region Östergötland, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lilliecreutz C, Soderstrom E, Ersson M, Bendtsen M, Brown V, Kaegi-Braun N, Linder R, Maddison R, Chisalita SI, Lof M. SPARK: an mHealth intervention for self-management and treatment of gestational diabetes mellitus in Sweden - protocol for a randomised controlled trial. BMJ Open. 2025 Mar 3;15(3):e089355. doi: 10.1136/bmjopen-2024-089355. PMID 40032379